CLINICAL TRIAL: NCT03437863
Title: Capitalizing on the Strengths of Persons With Rheumatoid Arthritis to Improve Health and Wellness
Brief Title: Feasibility of a Mobile Application to Support Reflection and Dialog About Strengths in People With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Elin Borosund, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015065
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Chronic Disease; Rheumatic Diseases
Keywords: self-management; health assets; Strengths; mHealth; Feasibility
MeSH Terms: conditions — Chronic Disease; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be recruited to a pre-post design study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application (Experimental): Participants recruited from a self-management course are asked to use (single time) a mobile application to support reflection of personal strengths. The participant borrows an Ipad and uses the application to 1) reflect and identify their strengths by reviewing a list of examples, 2) define personal goals, and 3) link strengths to goals.
  Interventions: Device: Mobile application

INTERVENTIONS:
Device: Mobile application — Use of a mobile application (on a borrowed device) with following features: 1) strengths reflection and identification, 2) summary of registered strengths, 3) defining goals, and 4) linking strengths to goals.

SUMMARY:
Self-management of chronic illness can be highly demanding and people need to mobilize their personal strengths in order to live well with their condition. A mobile application was designed in collaboration with people with chronic illness and health care providers with the aims to support awareness of patients' strengths and patient-provider dialogues that include strengths. The aim of the present study is to evaluate with mixed methods the perceived usefulness and usability of the application and potential effects of the application on patients.

DETAILED DESCRIPTION:
In this pre-post design pilot study participants will be recruited from self-management courses for people with rheumatic diseases. Before using the application participants will be asked to report their strengths in a written format. After using the mobile application to reflect on their strengths the participants will be interviewed about their experience of using the application and on the task of reflecting on their strengths. They will also be asked to fill out a questionnaire on perceived usefulness and user-friendliness. Before and after using the application the participants fill out questionnaires on emotions (Positive and Negative Affective Scale) and self-efficacy (The Arthritis Self-efficacy Scale). All interviews will be audio-taped and analyzed with a qualitative approach. Descriptive analysis will be applied for quantitative data.

ELIGIBILITY:
Setting 1:

Inclusion Criteria:

* Age of 18 years or older
* Can read and speak Norwegian language
* Diagnosed with a chronic condition
* Participating or having recently participated in a learning and mastery or an outpatient rehabilitation program

No exclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olöf B Kristjansdottir, PhD, Principal Investigator — Oslo University Hospital, Center for Shared Decision Making and Collaborative Care Research
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Application
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Application
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 50.0 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Perceived Usefulness of the Application
Description: Study-specific questions on perceived usefulness of the application
Time Frame: Within an hour after using the application
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Application
Number analyzed (Participants) | 12
Participants
  It was meaningful and relevant to use the app: Agree or strongly agree | 12
  It was meaningful and relevant to use the app: Disagree or strongly disagree | 0
  It was meaningful and relevant to use the app: Neutral | 0
  It was meaningful and relevant to use the app: Mssing | 0
  I became more aware of my own strengths by using the app: Agree or strongly agree | 9
  I became more aware of my own strengths by using the app: Disagree or strongly disagree | 1
  I became more aware of my own strengths by using the app: Neutral | 2
  I became more aware of my own strengths by using the app: Mssing | 0
  It was useful for me to see an overview of my own strengths: Agree or strongly agree | 10
  It was useful for me to see an overview of my own strengths: Disagree or strongly disagree | 0
  It was useful for me to see an overview of my own strengths: Neutral | 2
  It was useful for me to see an overview of my own strengths: Mssing | 0
  It was useful for me to be able to register a goal: Agree or strongly agree | 5
  It was useful for me to be able to register a goal: Disagree or strongly disagree | 2
  It was useful for me to be able to register a goal: Neutral | 4
  It was useful for me to be able to register a goal: Mssing | 1
  It was useful for me to be able to link the strengths to concrete goals: Agree or strongly agree | 6
  It was useful for me to be able to link the strengths to concrete goals: Disagree or strongly disagree | 0
  It was useful for me to be able to link the strengths to concrete goals: Neutral | 5
  It was useful for me to be able to link the strengths to concrete goals: Mssing | 1
  I liked the possibility to register my own notes: Agree or strongly agree | 7
  I liked the possibility to register my own notes: Disagree or strongly disagree | 0
  I liked the possibility to register my own notes: Neutral | 4
  I liked the possibility to register my own notes: Mssing | 1
  For me it would be relevant to share the overview of my strengths with my healthcare provider: Agree or strongly agree | 8
  For me it would be relevant to share the overview of my strengths with my healthcare provider: Disagree or strongly disagree | 0
  For me it would be relevant to share the overview of my strengths with my healthcare provider: Neutral | 4
  For me it would be relevant to share the overview of my strengths with my healthcare provider: Mssing | 0
  It was boring to use the app: Agree or strongly agree | 2
  It was boring to use the app: Disagree or strongly disagree | 9
  It was boring to use the app: Neutral | 1
  It was boring to use the app: Mssing | 0
  It was demanding for me to use the app: Agree or strongly agree | 1
  It was demanding for me to use the app: Disagree or strongly disagree | 11
  It was demanding for me to use the app: Neutral | 0
  It was demanding for me to use the app: Mssing | 0
  I would like to have the app on my own mobile devise: Agree or strongly agree | 7
  I would like to have the app on my own mobile devise: Disagree or strongly disagree | 2
  I would like to have the app on my own mobile devise: Neutral | 3
  I would like to have the app on my own mobile devise: Mssing | 0
  I would recommend the app to others in my situation: Agree or strongly agree | 9
  I would recommend the app to others in my situation: Disagree or strongly disagree | 0
  I would recommend the app to others in my situation: Neutral | 3
  I would recommend the app to others in my situation: Mssing | 0

2. Primary Outcome: The System Usability Scale
Description: This 10 item questionnaire measures usability. Each item has 5 response options with total score ranging from 0 to 100. Higher values represent a better outcome.
Time Frame: Within an hour after using the application
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Mobile Application
Number analyzed (Participants) | 12
score on a scale | 86.3 [70 to 100]

3. Secondary Outcome: The Positive and Negative Affect Schedule.
Description: This scale measures positive and negative affect with two subscales (positive affect and negative affect). Positive affect subscale scores can range from 10-50, with higher scores representing higher levels of positive affect. Negative affect subscale scores can range from 10-50, with lower scores representing lower levels of negative affect.
Time Frame: Pre-intervention and post-intervention, within an hour after using the application
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Mobile Application
Number analyzed (Participants) | 12
score on a scale
  Positive emotion sub scale (pre-intervention) | 34.0 [31.0 to 46.0]
  Positive emotion sub scale (post-intervention) | 35.0 [28.0 to 45.0]
  Negative emotion subscale (pre-intervention) | 12.0 [10.0 to 23.0]
  Negative emotion (post-intervention) | 11.0 [10.0 to 16.0]

4. Secondary Outcome: The Arthritis Self-efficacy Scale
Description: This scale measures self-efficacy with two subscales with 5 response options. The "pain" subscale has 5 items and a score range from 0 to 20. The "other symptoms" subscale has 6 items and a score range from 0 to 24. Higher scores equal higher levels of self-efficacy.
Time Frame: Pre-intervention and post-intervention, within an hour after using the application
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Mobile Application
Number analyzed (Participants) | 12
score on a scale
  Pain sub scale (pre-intervention) | 12.0 [5.0 to 16.0]
  Pain sub scale (post-intervention) | 14.0 [6.0 to 17.0]
  Other symptoms sub scale (pre-intervention) | 16.0 [8.0 to 22.0]
  Other symptoms subscale (post-intervention) | 17.0 [10.0 to 22.0]

ADVERSE EVENTS:
Time Frame: Within about 1 hour from testing the application.
Description: Observations.
Arm/Group | Mobile Application
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03437863/Prot_SAP_000.pdf